CLINICAL TRIAL: NCT00501969
Title: An Open-Label Extension to the Double-Blind SP515 (NCT00244387) Trial to Assess the Safety of Long-Term Treatment of Rotigotine in Subjects With Advanced-Stage Idiopathic Parkinson's Disease Who Are Not Well Controlled on L-Dopa
Brief Title: An Open-Label Extension Trial to Assess the Safety of Long-Term Treatment of Rotigotine in Advanced-Stage Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0516; 2004-000148-26 (EudraCT Number)
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Results first posted 2010-01-12 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2012-03

CONDITIONS: Advanced Stage Parkinson's Disease
Keywords: Rotigotine; Neupro®
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rotigotine (Experimental): Rotigotine
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Rotigotine trans-dermal patches once daily:
  20 cm2 (4 mg/24 hours); 30 cm2 (6 mg/24 hours); 40 cm2 (8 mg/24 hours) 50 cm2 (10 mg/24 hours) 60 cm2 (12 mg/24 hours) 70 cm2 (14 mg/24 hours) 80 cm2 (16 mg/24 hours)
  Other Names: Neupro®

SUMMARY:
The objective of this open-label extension is to assess the safety and tolerability of long-term treatment of the rotigotine patch in subjects with advanced-stage idiopathic Parkinson's disease

DETAILED DESCRIPTION:
This is the open-label extension to the randomized, double-blind, placebo-and active controlled SP515 (NCT00244387) trial that assessed the efficacy and safety and tolerability of the Rotigotine patch in subjects with advanced-stage idiopathic Parkinson's Disease that were not well-controlled on levodopa

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed four months of maintenance treatment in the SP515 (NCT00244387) double-blind trial

Exclusion Criteria:

* Subjects who had an ongoing serious adverse event from SP515 (NCT00244387) double-blind trial that was assessed as related to study medication

Min Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2004-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (53):
- Australia (5):
  - Bedford Park
  - Concord
  - Darlinghurst
  - East Gosford
  - Westmead
- Innsbruck, Austria
- Zagreb, Croatia
- Czechia (5):
  - Brno
  - Ostrava - Poruba
  - Pardubice
  - Pilsen
  - Prague
- Finland (2):
  - Oulu
  - Pori
- France (3):
  - Aix-en-Provence
  - Lille
  - Lyon
- Germany (2):
  - Aachen
  - Bochum
- Hungary (3):
  - Budapest
  - Miskolc
  - Pécs
- Israel (2):
  - Petah Tikva
  - Tel Aviv
- Italy (6):
  - Milan
  - Napoli
  - Padua
  - Pisa
  - Pozzilli
  - Roma
- New Zealand (3):
  - Auckland
  - Christchurch
  - Wellington
- Norway (4):
  - Bergen
  - Stavanger
  - Trondheim
  - Tønsberg
- Poland (6):
  - Gdansk
  - Krakow
  - Lublin
  - Mosina k/Poznania
  - Olsztyn
  - Warsaw
- South Africa (3):
  - Cape Town
  - Pretoria
  - Tygerberg
- Spain (3):
  - Barcelona
  - Donostia / San Sebastian
  - Madrid
- Stockholm, Sweden
- United Kingdom (3):
  - Blackpool
  - Glasgow
  - Sheffield

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An Open-Label Extension to the Double-Blind SP515 (NCT00244387) Trial to Assess the Safety of Long-Term Treatment of Rotigotine in Subjects with Advanced-Stage Idiopathic Parkinson's Disease who are not well controlled on L-Dopa from August 2004 to December 2008
Groups:
- Rotigotine: Optimal dosing for Rotigotine transdermal patches, once daily: Subjects can receive a dose up to 16 mg/24 hours.
Period: Overall Study
Arm/Group | Rotigotine
Started | 395
Completed | 189
Not Completed | 206
Not completed — Major Protocol Violation | 4
Not completed — Lack of Efficacy | 29
Not completed — Adverse Event | 76
Not completed — Unsatisfactory compliance of subject | 7
Not completed — Subject withdrew consent | 51
Not completed — Lost to Follow-up | 4
Not completed — Other: Tired Of Clinical Trial Process | 1
Not completed — Other: Sponsors Request | 10
Not completed — Other: Sponsor Termination at Site | 1
Not completed — Other: Sponsor Stopped Study | 12
Not completed — Other: Severe Dementia Unable Sign PIC | 1
Not completed — Other: Patients + Investigator Agreement | 1
Not completed — Other: Patient is Going to Have DBS | 1
Not completed — Other: Pat Pending Surgery for PD | 1
Not completed — Other: DX Changed - Parkinsons to PSNP | 1
Not completed — Other: As Required by Local EC | 2
Not completed — Other: Admin Request from the Sponsor | 3
Not completed — Other: Sponsor Termination/Commercial RX | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rotigotine
Number analyzed (Participants) | 395
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 183
  >=65 years | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144
  Male | 251
Region of Enrollment [Number; unit: participants]
  Finland | 8
  Spain | 35
  Austria | 6
  Israel | 22
  United Kingdom | 10
  Italy | 33
  France | 9
  Czech Republic | 50
  Hungary | 11
  Poland | 65
  Croatia | 27
  Australia | 30
  South Africa | 52
  Germany | 4
  Norway | 8
  New Zealand | 16
  Sweden | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Adverse Event During This Open-label Extension Study
Description: Adverse events are any untoward medical occurrences in a subject administered study treatment, whether or not these events are related to treatment.
Time Frame: five years
Population: Of the 395 subjects who entered the study, 395 are included in this summary based on the Safety Set (SS).
Measure: Number; unit: Subjects
Arm/Group | Rotigotine
Number analyzed (Participants) | 395
Subjects | 357

2. Secondary Outcome: Number of Subjects Who Withdrew From the Trial Due to an Adverse Event
Description: as for outcome 1
Time Frame: five years
Population: Of the 395 subjects who entered the study, 395 are included in this summary based on the Safety Set (SS).
Measure: Number; unit: Subjects
Arm/Group | Rotigotine
Number analyzed (Participants) | 395
Subjects | 76

3. Secondary Outcome: Mean Epworth Sleepiness Scale Score During the Open-label Extension
Description: The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. The total ESS score is the sum of 8 item-scores and can range between 0 and 24. The higher the score, the higher the person's level of daytime sleepiness.
Time Frame: Visit 13 (end of year 1), Visit 17 (end of year 2), Visit 21 (end of year 3), Visit 25(end of year 4)
Population: Of the 395 subjects who entered the study, 395 are included in this summary based on the Safety Set (SS). Last observation carried forward (LOCF) was utilized.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 395
Score on a scale
  Visit 13 (end of year 1) (n=377) | 7.4 (4.7)
  Visit 17 (end of year 2) (n=377) | 7.8 (5.1)
  Visit 21 (end of year 3) (n=377) | 8.0 (5.1)
  Visit 25 (end of year 4) (n=377) | 8.3 (5.2)

ADVERSE EVENTS:
Time Frame: Up to five years
Arm/Group | Rotigotine
Serious Adverse Events (participants affected / at risk) | 148/395
Other Adverse Events (participants affected / at risk) | 305/395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=395)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 4 (4)
Sick sinus syndrome (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 3 (3)
Cardiac arrest (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 1 (1)
Keratoconus (Eye disorders) | 1 (1)
Maculopathy (Eye disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1)
Periodontitis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 3 (3)
Application site reaction (General disorders) | 2 (2)
Gait disturbance (General disorders) | 2 (2)
Unevaluable event (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Implant site haematoma (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Transplant rejection (Immune system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 7 (8)
Bronchitis acute (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5)
Cellulitis (Infections and infestations) | 3 (3)
Arthritis infective (Infections and infestations) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Abscess (Infections and infestations) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Narcotic intoxication (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (5)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2)
Bursa disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Parkinson's disease (Nervous system disorders) | 18 (22)
Parkinsonism (Nervous system disorders) | 4 (5)
Cerebral haemorrhage (Nervous system disorders) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Loss of consciousness (Nervous system disorders) | 2 (2)
Radicular pain (Nervous system disorders) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (1)
Dyskinesia (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Sciatica (Nervous system disorders) | 2 (4)
Dementia (Nervous system disorders) | 1 (1)
Monoparesis (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Sudden onset of sleep (Nervous system disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 4 (4)
Hallucination, visual (Psychiatric disorders) | 4 (4)
Delirium (Psychiatric disorders) | 2 (2)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1)
Sleep attacks (Psychiatric disorders) | 1 (1)
Delusional disorder, persecutory type (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Pathological gambling (Psychiatric disorders) | 1 (2)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 6 (7)
Haematuria (Renal and urinary disorders) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Bladder disorder (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Prostatism (Reproductive system and breast disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep brain stimulation (Surgical and medical procedures) | 3 (3)
Knee arthroplasty (Surgical and medical procedures) | 3 (3)
Drug therapy changed (Surgical and medical procedures) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (1)
Spinal operation (Surgical and medical procedures) | 1 (1)
Open reduction of fracture (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Thrombophlebitis (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Cardiovascular insufficiency (Vascular disorders) | 1 (2)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (2)
Aortic aneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=395)
Nausea (Gastrointestinal disorders) | 54 (62)
Constipation (Gastrointestinal disorders) | 26 (29)
Application site erythema (General disorders) | 40 (45)
Application site pruritus (General disorders) | 38 (39)
Application site reaction (General disorders) | 29 (32)
Oedema peripheral (General disorders) | 33 (35)
Urinary tract infection (Infections and infestations) | 27 (46)
Fall (Injury, poisoning and procedural complications) | 61 (117)
Weight decreased (Investigations) | 43 (52)
Weight increased (Investigations) | 30 (32)
Back pain (Musculoskeletal and connective tissue disorders) | 48 (57)
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 (36)
Somnolence (Nervous system disorders) | 133 (170)
Dyskinesia (Nervous system disorders) | 55 (74)
Parkinson's disease (Nervous system disorders) | 44 (52)
Dizziness (Nervous system disorders) | 27 (31)
Headache (Nervous system disorders) | 27 (33)
Hallucination (Psychiatric disorders) | 32 (35)
Hallucination, visual (Psychiatric disorders) | 20 (27)
Insomnia (Psychiatric disorders) | 45 (52)
Depression (Psychiatric disorders) | 31 (33)
Abnormal dreams (Psychiatric disorders) | 20 (23)
Orthostatic hypotension (Vascular disorders) | 20 (21)
Hypertension (Vascular disorders) | 24 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.